CLINICAL TRIAL: NCT02645916
Title: Efficacy and Safety of Danggui-Sayuk-Ga-Osuyu-Saenggang-tang on Korean Patients With Cold Hypersensitivity in the Hands
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Sangji University Oriental Medical Hospital (Unknown); Semyung University Affiliated Oriental Medical Hospital (Other); Kyunghee University Medical Center (Other); Kyung Hee University Hospital at Gangdong (Other); DongGuk University (Other)
Responsible Party: Principal Investigator, Chan-Yong Jeon, PhD, KMD, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISEE_2015_DSGOST
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Cold Hypersensitivity
Keywords: Cold Hypersensitivity in the Hands; Korean medicine; DSGOST
MeSH Terms: conditions — Cold Hypersensitivity | interventions — DSGOST

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSGOST (Experimental): admission to Danggui-Sayuk-Ga-Osuyu-Saenggang-tang granule
  Interventions: Drug: Danggui-Sayuk-Ga-Osuyu-Saenggang-tang
- Placebo (Placebo Comparator): admission to placebo
  Interventions: Drug: Placebo: corn starch

INTERVENTIONS:
Drug: Danggui-Sayuk-Ga-Osuyu-Saenggang-tang — Usage: 3g, three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Other Names: DSGOST; Dangsanin Granule
  Arms: DSGOST
Drug: Placebo: corn starch — Usage: 3g three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Arms: Placebo

SUMMARY:
The Purpose of this trial is to investigate the efficacy and safety of Danggui-Sayuk-Ga-Osuyu-Saenggang-tang(DSGOST) on Korean Patients With Cold Hypersensitivity in the Hands

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 19 to 59 years have a complaint of CHH.
2. Patients must include at least one or more of the following symptoms:

   * Those who have the symptoms of CHH in normal temperature which most individuals feel no cold;
   * Those who have the symptoms of extremely cold hands in cold temperature exposure;
   * Those who are on the return to a warmer environment, the symptoms of cold hands is not completely rewarmed;
3. Those who have 4 cm or greater of VAS CHH score;
4. A thermal differences between the palm (PC8) and the upper arm (LU4) may be higher than 0.3℃;
5. Those who can comply with all study-related procedures, medications, and evaluations;
6. Given a written informed consent form.

Exclusion Criteria:

We will exclude patients who have taken

1. Patients with calcium antagonists or beta-blockers with the purpose of treating CHH;
2. Those who have one or more finger gangrene or ulceration;
3. Those who are diagnosed by hypothyroidism or currently medicated to thyroid drugs;
4. Those who are diagnosed by autoimmune disease or have a positive ANA test result;
5. Those who are diagnosed by carpal tunnel syndrome or have a positive Tinel and Phalen's tests;
6. Those who are diagnosed with cervical disc herniation or (malignant) tumor disease;
7. Those who are diagnosed with diabetes;
8. Those who are currently medicated to drugs that may affect to CHH symptoms, such as anticoagulants etc;
9. Those who have moderate level of liver dysfunction (each of AST, ALT greater than 100 IU/L) or kidney dysfunction (Cr 2.0mg/dL);
10. Those who do not (cannot) abide by treatment and follow up due to the mental illness such as behavior disorder, depression, anxiety neurosis, schizophrenia, or serious mental illness;
11. Those who are Diagnosed with moderate anemia and hematologic disorders (adult non-pregnant women hemoglobin (Hgb) level less than 7g/dL, hematocrit (Hct) level less than 26%, white blood cell (WBC) level greater than 11,000/mm3);
12. Those whose systolic blood pressure (SBP) 180mmHg or diastolic blood pressure (DBP) is greater than 100 mmHg based on average value of at least 2 measurements;
13. Those who are suspected arrhythmia that showing up on ECG, or diagnosed by heart diseases, such as, ischemic heart disease and so on;
14. Those who are addicted to alcohol or drugs;
15. Those who are pregnant (positive urine-HCG) or lactating or have the chances of pregnancy;
16. Those who are currently participated in other clinical trials;
17. Those who are able to understand and speak Korean;
18. Those who are judged to be inappropriate for the clinical study by the researchers.

Ages: 19 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in visual analogue scale | At baseline, week 2, 4, 6

SECONDARY OUTCOMES:
Changes from baseline in body temperature | At baseline, week 2, 4, 6
Changes from baseline in clinical global impression(CGI) | At baseline, week 2, 4, 6
Changes from baseline in WHOQoL-BREF | At baseline, week 2, 4, 6
Changes from baseline in cold stress test | At baseline, week 6
  similar to the cold stimulation test

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University, Gil Oriental Medicine Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ko Y, Go HY, Cho YY, Shin JH, Kim TH, Choi DJ, Lee JM, Jang JB, Song YK, Ko SG, Sun SH, Jeon CY. The efficacy and safety of Danggui-Sayuk-Ga-Osuyu-Saenggang-tang on Korean patients with cold hypersensitivity in the hands: study protocol for a pilot, double-blind, randomized, placebo-controlled, parallel-group clinical trial. Trials. 2017 Jun 8;18(1):268. doi: 10.1186/s13063-017-2002-8. PMID 28595610